CLINICAL TRIAL: NCT02086617
Title: Screening of Abdominal Aortic Aneurysms Among Men With Coronary Artery Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: North Karelia Central Hospital (Other)
Responsible Party: Sponsor
Purpose: Screening
Other Study IDs: AAA-CAD-04
Record Dates: First submitted 2014-03-11; First posted 2014-03-13 (Estimated); Last update posted 2014-06-26 (Estimated); Status verified 2014-06

CONDITIONS: Abdominal Aortic Aneurysm
MeSH Terms: conditions — Aortic Aneurysm, Abdominal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ultrasound of aorta (Other)
  Interventions: Other: ultrasound of aorta

INTERVENTIONS:
Other: ultrasound of aorta

SUMMARY:
The purpose of this study is to investigate prevalence of abdominal aortic aneurysms (AAA) among male patients with coronary artery disease (CAD). Secondary purpose is to document cost-effectiveness of ultrasound screening of AAA in selected population.

Ethiology of AAA is known to be common with atherosclerotic arterial diseases, and on the basis of our previous studies (ClinicalTrials.gov ID CAD-AAA-02) the prevalence of AAA seems to be higher in CAD population than unselected male population. This leads to hypothesis that selective screening of these patients (for AAA) could be cost-efficient and life saving option for detecting AAAs before rupture.

Study will be carried out as a single-center prospective screening study. Patients will be selected for this study on basis of their ICD 10 diagnose codes in North Carelian patient information system. Inclusion criteria will be any kind of atherosclerotic heart disease (ICD10 codes I20-I25). Criteria for exclusion are malignant disease, already diagnosed or treated AAA and failure to give informed consent.

800 patient records that meet the inclusion criteria will be reviewed for eligibility. Invitations for screening will be sent for 600 patients with intention to have at least 400 patients screened. Screening will be done by verified sonographers in designated screening appointments.

ELIGIBILITY:
Inclusion Criteria:

* Male patients with coronary artery disease

Exclusion Criteria:

* Already diagnosed or treated abdominal aortic aneurysm
* Patient's denial to participate
* Malignant disease

Min Age: 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2014-03; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Maximum diameter (mm) of abdominal aorta (outer-to-outer wall) in ultrasound | Upon screening (AAA-screening appointment, 10 minutes per patient)

CONTACTS AND LOCATIONS:
Locations (1):
- North Carelia Central Hospital, Joensuu, Pohjois-Karjala, Finland